CLINICAL TRIAL: NCT05204628
Title: Randomized Multicenter Phase III Open-Label Study to Evaluate and Compare the Efficacy and Safety of XZP-3621 Versus Crizotinib in Chinese Patients With Treatment-Naive Anaplastic Lymphoma Kinase-Positive Advanced Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate and Compare the Efficacy and Safety of XZP-3621 Versus Crizotinib
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XZP-3621-3001
Record Dates: First submitted 2021-12-20; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: XZP-3621; Crizotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XZP-3621 (Experimental): Participants will receive XZP-3621 tablets orally at a dose of 500 mg QD with food until disease progression, unacceptable toxicity withdrawal of consent, or death, whichever occurred first.
  Interventions: Drug: XZP-3621
- Crizotinib (Active Comparator): Participants will receive crizotinib capsules orally at a dose of 250 mg BID with or without food until disease progression, unacceptable toxicity withdrawal of consent, or death, whichever occurred first.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: XZP-3621 — XZP-3621 tablets will be administered orally at a dose of 500 mg QD until disease progression, unacceptable toxicity withdrawal of consent, or death, whichever occurred first.
  Arms: XZP-3621
Drug: Crizotinib — Crizotinib capsules will be administered orally at a dose of 250 mg BID until disease progression, unacceptable toxicity withdrawal of consent, or death, whichever occurred first.
  Arms: Crizotinib

SUMMARY:
This randomized, multicenter, Phase III, open-label study will evaluate the efficacy and safety of XZP-3621 versus crizotinib and to evaluate the pharmacokinetics of XZP-3621 in Chinese participants with treatment-naive ALK-positive advanced NSCLC. Participants will be randomized 1:1 into one of the two treatment groups to receive either XZP-3621 (500 milligrams [mg] once daily [QD]) or crizotinib (250 mg BID) orally, respectively.

DETAILED DESCRIPTION:
This is a randomized, active controlled, multicenter Phase III open-label study in patients with treatment-naive ALK-positive advanced NSCLC. Patients will be randomized 1:1 into one of the two treatment arms to receive either XZP-3621 or crizotinib. The primary endpoint of the study is investigator-assessed PFS.

Central randomization will be performed via a web-based response system using the following stratification factors: chemotherapy (yes vs. no) and CNS metastases at baseline (yes vs. no).

The experimental arm will receive XZP-3621 at 500 mg orally once daily (QD), taken with food. The control arm will receive crizotinib at 250 mg orally BID, taken with or without food.

Patients will be treated until disease progression, unacceptable toxicity, withdrawal of consent, or death. After disease progression (as per RECIST v1.1), patients should discontinue the study medication. After disease progression, patients will be treated at the discretion of the investigator according to local practice. Information regarding the nature and the duration of subsequent therapies will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18-75 years-of-age;
2. Patients with Histologically or cytologically confirmed diagnosis of advanced or recurrent (Stage IIIB and IIIC not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC that is ALK-positive where ALK status is determined by the NMPA-approved (for use in China) Ventana (D5F3) immunohistochemistry (IHC) test or FISH or PCR or NGS, Sufficient tumor tissue available to perform ALK status is required if not determined.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 2;
4. Life expectancy of at least 12 weeks;
5. Ability to swallow and retain oral medication;
6. Adequate organ system function, defined as follows:

   1. Absolute neutrophil count (ANC) ≥1.5 x 109/L; Platelets ≥100 x 109/L; Hemoglobin ≥9 g/dL (≥90 g/L)
   2. Total bilirubin ≤1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 *ULN if no liver involvement or ≤5 * ULN with liver involvement.
   3. Creatinine < 1.5 *ULN. If >1.5 * ULN, patient may still be eligible if calculated creatinine clearance >50 mL/min (0.83mL/s) as calculated by the Cockcroft-Gault method.
7. No prior systemic treatment for advanced or recurrent NSCLC (Stage IIIB and IIIC not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC
8. Tumor Requirements: At least 1 extracranial measurable target lesion per RECIST v. 1.1 that has not been previously irradiated.
9. Serum pregnancy test (for females of childbearing potential) negative at screening.
10. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Patients with a previous malignancy within the past 3 years are excluded (other than curatively treated basal cell carcinoma of the skin, early gastrointestinal (GI) cancer by endoscopic resection, in situ carcinoma of the cervix, or any cured cancer that is considered to have no impact in PFS and OS for the current NSCLC).
2. Any GI disorder that may affect absorption of oral medications, such as mal-absorption syndrome or status post-major bowel resection ;
3. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV) or hepatitis C virus (HCV) (eg, in case of known HBsAg or HCV antibody positivity), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness;
4. Clinically significant vascular (both arterial and venous) and non-vascular cardiac conditions, (active or within 3 months prior to enrollment), which may include, but are not limited to:

   1. Arterial disease such as cerebral vascular accident/stroke (including Transient Ischemic Attack -TIA), myocardial infarction, unstable angina;
   2. Venous diseases such as cerebral venous thrombosis, symptomatic pulmonary embolism;
   3. Non-vascular cardiac disease such as congestive heart failure (New York Heart Association Classification Class ≥ II), second-degree or third-degree AV block (unless paced) or any AV block with PR >220 msec; or ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, etc.), machine-read Electrocardiogram (ECG) with QTc >470 msec, or congenital long QT syndrome;
5. Patients with predisposing characteristics for acute pancreatitis according to investigator judgment (eg, uncontrolled hyperglycemia, current gallstone disease) in the last month prior to randomization;
6. History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis;
7. Concurrent use of known strong CYP3A4 inhibitors and inducers (consult the sponsor if in doubt whether a food or a drug falls into any of the above categories) within 7 days prior to the first dose of XZP-3621 or crizotinib.
8. Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation;
9. Pregnant female patients; breastfeeding female patients;
10. History of organ transplant;
11. Co-administration of anti-cancer therapies other than those administered in this study;
12. Baseline QTc>470ms ;
13. History of hypersensitivity to any of the additives in the XZP-3621 or crizotinib drug formulation;
14. Any psychological condition that potentially hampers compliance with the study protocol requirements or follow-up procedures; this condition should be discussed with the participant before study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2022-02-07 (Estimated); Primary Completion 2025-05-07 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of randomization to the date of the first documented disease progression or death, whichever occurred first (up to overall period of approximately 30 months)
  PFS was defined as the time (in months) from randomization to the first documentation of disease progression, as determined by investigators using Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 or to death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of randomization to the date of the first documented disease progression or death, whichever occurred first (up to overall period of approximately 30 months).
  PFS was defined as the time (in months) from randomization to the first documentation of disease progression, as Determined by Blind Independent Central Review(BICR)Using RECISTv1.1., or to death from any cause, whichever occurred first.
Overall Survival (OS) | From randomization until death (up to approximately 30 months).
  OS defined as time from date of randomization to date of death due to any cause, as Determined by the investigator and Blind Independent Central Review (BICR) Using RECISTv1.1
Overall Response Rate (ORR) | From randomization until death (up to approximately 30 months)
  ORR defined as the proportion of patients with a best overall response defined as Complete Response (CR) or Partial Response (PR) as evaluated by Blinded Independent Central Review (BICR) and by investigator assessment per RECIST 1.1
Duration of Response (DOR) | From randomization until death (up to approximately 30 months)
  DOR defined as the time from date of first documented CR or PR to date of first documented disease progression or death due to any cause
Disease Control Rate (DCR) | Baseline, Week 8, thereafter every 8 weeks until disease progression, death or withdrawal from the study (up to overall period of approximately 30 months)
  DCR defined as the proportion of patients with best overall response of CR, PR, or Stable Disease (SD)
Intracranial Objective Response Rate (IC-ORR) | Baseline, Week 8, thereafter every 8 weeks until disease progression, death or withdrawal from the study (up to overall period of approximately 30 months)
  IC-ORR as Determined by BICR and investigator Using Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
Intracranial Duration of Response (IC-DoR) | Baseline, Week 8, thereafter every 8 weeks until disease progression, death or withdrawal from the study (up to overall period of approximately 30 months)
  IC-ORR as Determined by BICR and investigator Using Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
Area Under the Plasma Concentration-time Curve (AUC) of XZP-3621 and Its Metabolite | Pre-dose (within 1 hour before XZP-3621), 4 hours post-dose at first dosing day and Week 4; Pre-dose (within 1 hour) at Week 8,12,16 (up to 4 months)
  AUC was collected for both XZP-3621 and its major metabolite, and was based on their concentrations in plasma over time.
Maximum Plasma Concentration Observed (Cmax) of XZP-3621 and Its Metabolite | Pre-dose (within 1 hour before XZP-3621), 4 hours post-dose at first dosing day and Week 4; Pre-dose (within 1 hour) at Week 8,12,16 (up to 4 months)
  Cmax was collected for both XZP-3621 and its major metabolite, and was based on their concentrations in plasma over time.
Time to Deterioration by EORTC Quality of Life Questionnaire Lung Cancer Module 13 (LC13) | Baseline, Week 4, thereafter every 4 weeks until disease progression, death or withdrawal from the study and 2 weeks after permanent discontinuation (up to overall period of approximately 30 months)
  The EORTC QLQ-LC13 module generated one multiple-item scale score assessing dyspnea and a series of single item scores assessing chest pain, arm/shoulder pain, pain in other parts, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All the scales and single-item scores were linearly transformed so that each score ranged from 0 to 100. A higher score on the global health and functioning subscales is indicative of better functioning. Confirmed clinically meaningful deterioration in lung cancer symptoms is defined as a >or=10-point increase from baseline in a symptom score that must be held for at least two consecutive assessments or an initial >or=10-point increase above baseline followed by death within 5 weeks from the last assessment.
Change From Baseline in Global Health Status/Quality of Life as Assessed by EORTC QLQ-C30 | Baseline, Week 4, thereafter every 4 weeks until disease progression, death or withdrawal from the study and 4 weeks after permanent discontinuation (up to overall period of approximately 30 months)
  HRQoL: perceived quality of participant's life, includes self-reported multidimensional measures of physical and mental health. Patient-reported symptoms (PROs) and HRQoL will be collected by administering the european organisation for research and treatment of cancer (EORTC) quality of life (QLQ)-C30 questionnaire. EORTC-QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status/QOL scale. The 30 items have 4 response levels (not at all, a little, quite a bit, and very much), with 2 questions relying on a 7-point numeric rating scale. Raw scores are converted into overall score ranging from 0 to 100, where lower scores indicate better QOL. A negative change from Baseline indicates improvement.
Percentage of Participants with Non-serious Adverse Events and Serious Adverse Events | Up to overall period of approximately 30 months
  Percentage of Participants with Non-serious, Adverse Events and Serious Adverse Events. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, MD, Principal Investigator — Jilin Province Cancer Hospital
Locations (1):
- Jilin Province Cancer Hospital, Changchun, Jilin, China